CLINICAL TRIAL: NCT03548896
Title: Dimensional Changes Following Ridge Augmentation of the Buccal Wall in Dehiscence Sockets: a Randomized-controlled Clinical Trial.
Brief Title: Ridge Regeneration in Three Wall Sockets
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Pedro Diz Iglesias, Principal investigator, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER 2016-02
Record Dates: First submitted 2018-01-28; First posted 2018-06-07 (Actual); Last update posted 2018-07-10 (Actual); Status verified 2018-07

CONDITIONS: Dental Implant; Socket Preservation
Keywords: implant

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dental Implants (Experimental): Dental implants Titanium SLA treated surface of different dimensions according to the specific needs of the patient
  Interventions: Procedure: Post extraction socket
- Resorbable membrane (Experimental): Resorbable membrane Cross link collagen membrane from porcine animal with a measure of 15 x 25 mm
  Interventions: Procedure: Post extraction socket
- Allograft (Experimental): Allograft Bone from human source that is administered in a dosage of 1 cc per patient
  Interventions: Procedure: Post extraction socket

INTERVENTIONS:
Procedure: Post extraction socket — **Dental implant will be placed 3 months after tooth extraction

SUMMARY:
There is limited data regarding socket preservation in three wall defects and no enough evidence of implant placement in previously regenerated area with allograft.

The aim of this randomized controlled clinical trial is to analyze and compare dimensional changes in extractions sites with buccal bone defects > 5 mm left untreated (simultaneous regeneration during implant placement) or treated using a mineralized allograft.

DETAILED DESCRIPTION:
1. Introduction:

   The alveolar process is tooth dependent and once a single tooth is extracted, the architecture of the socket undergoes dimensional changes hindering the prosthetic rehabilitation at the edentulous crest which demands a posterior guided bone regeneration (GBR). Studies in dogs described the main changes happened after tooth extraction (1,2); the blood forms a clot at the wound site which is replaced by a connective tissue matrix: after 1 month the woven bone fills the extraction socket; subsequently the woven bone undergoes osteoclastic resorption which leads to a maturation of the recently formed bone, gradually replaced with lamellar and bone marrow. Such events were clinically evaluated in several studies with an average of loss in width (3.5-4mm) (3). Bone resorption in height is correlated to the plate thickness; thin-wall phenotypes (<1mm) have a median vertical bone loss of 7.5mm in the central risk zone (4). Moreover, at the aesthetic zone, this narrow crest makes more difficult the adequate implant placement (5), then functional and esthetic complications can be expected.

   The fresh socket in the esthetic zone represents a challenge for the clinician and immediate implant placement (type I) is associated with a high risk of mucosal

   recessions. Moreover, the absence of the buccal plate increases the risk (6). Early implant placement (type II) described by Buser et al. (7) reported long term excellent esthetic results and this technique is compatible with alveolar ridge preservation.

   Alveolar ridge preservation is a widely used technique immediately after tooth extraction to minimize the alveolar resorption, to accelerate the bone formation and to improve the prosthetic restoration with an implant placed on a tridimensional way. Different biomaterials were used: autografts (8), allografts (9), xenografts (10,11), alloplasts (11,12) with or without barrier membranes. In all of them, less bone resorption was drawn with respect to natural healing; however, such techniques do not prevent physiologic bone resorption but limit it, improving the expected results in absence of preservation (13). Comparing the healing time with different biomaterials, mineralized bone allograft demonstrated similar results in the amount of new bone growth at 3 and 6 months after extraction (14) allowing the reentry before.

   In many cases, it is reported the absence of the buccal bone plate after tooth extraction; according to Chappuis et al. 2013 (4), at the anterior maxilla, central wall thickness has less than 1 mm in approximately 69% of the cases, increasing the risk of a resorption after healed or even it may disappear after tooth extraction due to the lack of consistency which affects aesthetics negatively.

   The bone remodeling not only happens among the three first millimeters (mm) as previously reported (2) and a primate model clearly demonstrated that the bone remodeling was not limited to the crestal 3-mm zone and extended up to 6 mm below the alveolar crest, where a mean volumetric bone loss of 30% and 45% at 6 and 12 weeks in intact sockets while more pronounced bone loss with 60 and 86% volumetric bone loss in the 0-3 mm zone, respectively, in the untreated dehiscence group and the use of biomaterials in combination with a membrane reduces the volumetric bone loss up to 25% (15).

   There is limited data regarding the effect of ridge preservation in 3 bone wall defects sockets. Some studies allowed partial bone wall (16-19), while only five studies have investigated the effect of alveolar ridge preservation on buccal wall defects (20-23). Alloplastic materials have evidenced adequate outcomes regarding ridge width maintenance requiring posterior guided bone regeneration at the implant surgery in a

   few cases (27,8%) (24) or no regeneration at two months post preservation (22).
2. Background:

   Dehiscence-type defect associated with the extraction socket still presents a problem if an implant is desired in such site. Recently published study has reported the necessity of posterior guided bone regeneration at the reentry for implant placement in 50% previously preserved ridges when using xenograft (23). No data regarding the effect on ridge preservation dehiscences is available using a mineralized allograft and membrane, and if it has benefits compared to the conventional guided bone regeneration at the implant placement.

   A recent systematic review recommends further research on ridge preservation assessing the integrity/absence of the buccal plate in the dimensional changes and long term evaluation of bone levels after implant placed in alveolar sockets previously treated with alveolar ridge preservation using standardized radiographs taken at specific period of times (25). Furthermore, the soft tissue volume stability is of great importance in a esthetic high risk zone (26) which was not reported in any previous study. Therefore, the aim of this randomized controlled clinical trial is to analyze and compare dimensional changes in extractions sites with buccal bone defects more than 5 mm left untreated or treated using a mineralized allograft.
3. Objectives:

   3.1 General objective

   To compare the dimensional changes in bone and soft tissues happened after tooth extraction in alveolus with dehiscences when using a mineral allograft and resorbable membrane (test group) or natural healing (control group) at 3 months.

   3.2 Specific objectives

   3.2.1 To compare bone changes in width and height from the baseline (immediately after tooth extraction) to the implant placement stage at 3 months, and at 12 months after tooth extraction between test and control groups.

   3.2.2 To compare marginal bone loss around implants, from the baseline (time of implant placement) to the second-stage surgery, at the prosthetic loading, and at 12 months after tooth extraction between test and control groups.

   3.2.3 To compare the facial soft tissue level at the baseline (immediately before tooth extraction) and at 3 months, at the second stage implant surgery, at the prosthetic loading, and at 12 months after tooth extraction between test and control groups.

   3.2.4 To compare volumetric changes at baseline, at 3 months (previous implant placement), at the second stage implant surgery, at the prosthetic loading, and at 12 months after tooth extraction between test and control groups.

   3.2.5 To compare the width of keratinized tissue at the baseline, at 3 months, before the second implant surgery, at the prosthetic loading, and at 12 months after tooth extraction between test and control groups.

   3.2.6 To compare the pink esthetic score at the end of the evaluation between test and control group.
4. Hypothesis:

   4.1 Null hypothesis
   * Ho1. Dimensional changes are greater in the test group than in the control group.
   * Ho2. Bone changes in width and height are greater in the test group than in the control group.
   * Ho3. Marginal bone loss around implants are greater in the test group than in the control group.
   * Ho4. The facial soft tissue level is worse maintained in the test group than in the control group.
   * Ho5. There are more volumetric changes in the soft tissues in the test group than in the control group.
   * H06. The width of the keratinized tissue is lower in the test group than in the control group.
   * H07. The pink esthetic score is fewer in the test group than in the control group.

   4.2 Alternative hypothesis
   * H11. Dimensional changes are lower in the test group than in the control group.
   * H12. Bone changes in width and height are lower in the test group than in the control group.
   * H13. Marginal bone loss around implants are greater in the test group than in the control group.
   * H14. The facial soft tissue level is better maintained in the test group than in the control group.
   * H15. There are less volumetric changes in the test group than in the control group.
   * H16. The width of the keratinized tissue is greater in the test group than in the control group.
   * H17. The pink esthetic score is higher in the test group than in the control group.
5. Material AND Methods:

   5.1 Study design

   This is a randomized controlled clinical trial with a 1-year follow-up. The recruitment of the patients will start on February 2016

   5.2 Setting of the study

   The study will be performed at the Universitat Internacional de Catalunya (UIC). Subjects will be recruited consecutively from the Department of Periodontology.

   5.3 Study population

   Patients referred to Department of Periodontology for treatment of periodontal diseases and who meet the inclusion criteria will be included in the study. Those with periodontal disease will be included in the study after periodontal treatment. Patients will be recruited consecutively. Furthermore, all study subjects will provide written informed consent before participating in the study. The study will be performed following the principles outlined in the Declaration of Helsinki (revised, amended, and clarified in 2013).

   5.4 Study procedures

   5.4.1 Screening examination

   Two calibrated investigators will evaluate and enroll the patients (P.D. and C.V.).

   The clinicians will review with the patient the Information and Medication History Forms and record the information. Patients will also be advised of their role in this study and asked to sign an informed consent. No patient will be admitted to the study until the

   informed consent form is signed. After giving consent, patients will undergo an oral pathology examination. After completion of the oral pathology exam, patients will undergo a full-mouth manual probing using a periodontal probe PCP-UNC 15 (HuFriedy, Rockwell St, Chicago, IL) to determine their periodontal status and, if needed, a full-mouth periapical radiographic examination.

   To take part in this study, one maxillary anterior tooth (from second premolar to second premolar) must show an absence of > 5mm of the buccal plate, measured with the periodontal probe PCP-UNC 15 (HuFriedy, Rockwell St, Chicago, IL) from the theoretical position of the alveolar crest.

   5.4.2 Study groups

   Patients will be randomly assigned to Test (n=14) or Control (n=14) groups using opaque envelopes after obtaining an automatic randomization list (generated with a software).
   * Control group (CG): after tooth extraction, a blood clot will be allowed to form in the alveolar defect. Augmentation of the buccal wall will be performed following socket healing, at the time of implant placement.
   * Test group (TG): after tooth extraction, the alveolar defect will be treated with mineralized allograft in combination with a resorbable collagen membrane.

   5.4.3 Therapeutic stages

   5.4.3.1 First part of the treatment protocol (alveolar ridge preservation OR natural healing of the socket)

   A) Hygienic phase

   All patients will receive presurgical therapy, which included oral hygiene instructions, a session of prophylaxis, and any periodontal treatment necessary to provide an oral environment more favorable to wound healing.

   B) Surgical phase

   B.1) Tooth extraction (T0)

   After initial therapy, the patient will be scheduled for tooth extraction. Surgical procedure will be carried out by second and third year residents of the Master of Periodontology and supervised by the same clinical instructor (C.V.). An alginate impression will be taken before the surgical procedure as baseline to measure the volumetric changes.

   Prior to the tooth extraction, patients will be instructed to rinse with 0.12% clorhexidine gluconate for 1 minute before induction of local anaesthesia (40 mgr.

   articaine, 0,01ml epinephrine). Pre-surgical medications will not be provided.

   Regarding the tooth extraction, all patients will be treated with the same surgical technique. The teeth will be extracted using a flapless, minimally invasive technique. A periodontal probe PCP-UNC 15 (HuFriedy, Rockwell St, Chicago, IL) will be used to measure the vertical distance (VD) between the buccal gingival margin and the bone wall. Periotomes will be used around each single tooth in order to prevent damage or full fracture of the facial bone wall. The extraction socket will be thoroughly curetted and irrigated with sterile saline solution.

   After extraction, all patients will undergo CT imaging (cone-beam computed tomography, CBCT). This will be used as baseline to measure the bone profile. All CT examinations will be carried out using the same cone-beam instrument. Afterwards, the randomization envelope will be opened and the sites will be allocated to test (regenerative procedure) or control (natural healing) groups.

   Subsequently, in the test group, extraction sockets will be filled with a mineralized allograft (OSTEOpureTM) placed, layer-by-layer, gently pressed to the extraction socket. A trimmed collagen membrane (Ossix Plus, Datum Dental) will be

   used to completely cover the socket; thus, extending 2-3 mm onto the alveolar defect without any further fixation. The soft tissues will be only undermined, and no

   releasing incisions will be performed. The collagen membrane will be left intentionally exposed to the oral cavity. On the contrary, in the control group, the post extraction alveolus will be filled with a collagen sponge (Octocolagen). Single interrupted non-resorbable polytetrafluoroethylene (PTFE) monofilament sutures (4-0 Cytoplast; Osteogenics Biomedical INC., Lubbock, TX, USA) will be used in both groups. Finally, a custom-

   made provisional fixed partial denture without tooth preparation of the adjacent teeth (FPD) included an ovate pontic to stabilize the graft material (in the test group) and support buccal soft tissues.

   Due to the nature of the study design, neither the patient nor the surgeon will be blinded.

   B.1.1) Post-surgical instructions

   Post-surgical instructions will be given to patients. A normal oral hygiene will be performed except in the surgical area, which will not be brushed until the suture is removed. After surgery, in the test group, amoxicillin 500 mg every 8 hours will be prescribed for the following 7 days (clindamycin 300 mg every 6 hours will be prescribed to penicillin-allergic patients). In order to control discomfort and swelling, non-steroidal anti-inflammatory treatment (600 mg ibuprofen every 8 hours for 4 days) will be administered to both groups. Ice packs will be used for 24 h and all subjects will be prescribed 0.12% chlorhexidine mouthrinse twice daily for 14 days for chemical plaque control.

   B.1.2) Evaluation visits

   After a healing period of 14 days, sutures will be removed. Patients will be observed monthly to control adequate tissue healing and after a 3-month healing period will be scheduled for re-entry and implant placement. A second alginate impression will be taken before implant placement for the volumetric analysis. A CBCT scan will be obtained before implant installation for treatment planning.

   5.4.3.2 Second part of the treatment protocol (implant placement and prosthetic rehabilitation)

   A) Implant placement (T1)

   Following the application of local anaesthesia (40 mgr. articaine, 0,01ml epinephrine), a crestal incision will be performed. Implant placement will be performed by second and third year residents and supervised by the same clinical instructor (J.N.). Buccal and lingual mucoperiosteal flaps will be carefully reflected and any soft tissue will be removed. Osteotomies will be prepared and dental implants will be placed according to

   manufacturer's recommendations in a prosthetically ideal position. After implant placement, the presence of a peri-implant bone defect will be evaluated; augmentation procedures will be considered necessary to treat the residual peri-implant bone defect. The regenerative procedure will be performed with the use of mineralized allograft (OSTEOpureTM) covered by a collagen membrane (Ossix Plus, Datum

   Dental). Periosteal releasing incisions will be made to the surgical sites to allow for tension-free coronal advancement of the flaps with complete closure of the sites. After closure screw insertion, the incisions will be carefully closed with horizontal mattress sutures as well as single interrupted non-resorbable polytetrafluoroethylene (PTFE) monofilament sutures (4-0 Cytoplast; Osteogenics Biomedical INC., Lubbock, TX, USA). Patients will receive the same drug regime as prescribed after the first surgical phase (i.e. regenerative procedure after tooth extraction). An intra-oral periapical radiograph will be taken with a long cone paralleling technique (7mA-60kV/20ms). A radiographic bite block will be used in order to provide reproducible measurements at each examination time point. The temporary prosthetic restoration used at the first surgical step will be applied.

   B) Second-stage surgery and subepithelial connective tissue graft (T2)

   Four months after implant placement, a second-stage implant surgery will be performed. An alginate impression will be taken before the surgical procedure for the volumetric analysis. Under infiltrative local anesthesia, a midcrestal incision will be made to the dental implant region and the mucosa will be raised with a tunneling instrument until the cover screw is reached. After removing the cover screws, healing abutments will be placed. A subepithelial connective tissue graft (SCTG)

   from the tuberosity will be obtained. A double incision using double-bladed knife separated by 1.5 mm will be made from the distal of the terminal tooth. A second incision joining the first one will be made perpendicular at a distal part. The donor area will be

   sutured and the SCTG will be de-epithelized and the required dimensions (10mm height, 12mm length, and 1.5mm thick) checked. Finally, the SCTG will be placed under the flap and stabilized with resorbable sutures. The buccal flap will be mobilized and wound closure will be achieved with a non-resorbable suture. The postoperative regimen and medication will be the same as after the implantation but no antibiotics will be administered. An intra-oral periapical radiograph will be taken and two weeks later the sutures will be removed.

   C) Prosthetic loading (T3)

   After 6 weeks of second-stage surgery, a fourth alginate impression will be taken before starting the prosthetic restoration. At the end of this stage (T3), a periapical radiograph will be taken. Patients will be subsequently enrolled onto an oral hygiene program with a recall visit every 3 months.

   D) Follow-up (T4)

   The patients will be followed up for 1 year after tooth extraction and a CBCT and a periapical radiograph will be performed to assess the buccolingual width changes and the interproximal marginal bone loss, respectively, in each group. Furthermore, the pink esthetic score (PES) according to Fürhauser et al. (26) will be assessed by the same calibrated examiner (C.V.). Finally, a fifth alginate impression and a CBCT scan will be taken at the end of the follow-up period.

   5.5 Data collection

   A guidebook will be prepared to standardize procedures throughout the protocol, step by step, for all questionnaires and evidence collection. The data will be transferred to a computerized database.

   5.5.1 Anthropometric and sociodemographic data

   An interview will be conducted to obtain information regarding age, race, gender, medical history, medication, and health behaviour (smoking habits). Smoking behaviour will be specified as 3 categories: never smoker, former smoker,

   or current smoker (light smokers: < 10 cigarettes/day). Patients will be asked about their tobacco smoke exposure in terms of consumption (i.e. the number of cigarettes consumed per day); duration (i.e. the number of years of smoking); and life-time exposure (i.e. the accumulated exposure as formed by the product of consumption and duration: cigarette-years). In case of former smokers, patients will be asked about the smoke-free time following cessation.

   5.5.2 Clinical parameters

   The following clinical parameters will be evaluated by one examiner (P.D.) using a manual periodontal probe PCP-UNC 15 (HuFriedy, Rockwell St, Chicago, IL) rounded to the nearest 0.5 mm.
   * Visible plaque index (VPI) (28) will be recorded at six sites per tooth (excluding third molars) at baseline (T0) and at T1, T2, T3, and T4 using a 0-1 measure, where 0 indicates no visible plaque and 1 the presence of dental plaque. The number of positive sites will be recorded and then expressed as a percentage of the numbers of sites examined (full-mouth plaque score).
   * Modified Plaque Index (mPlI) (29) will be recorded at four aspects (mesial, distal, buccal, and lingual) around each implant at T3 and T4:

     * Score 0: No detection of plaque
     * Score 1: Plaque only recognized by running a probe across the smooth marginal surface of the implant. Implants covered by titanium spray in this area always score 1.
     * Score 2: Plaque can be seen by the naked eye.
     * Score 3: Abundance of soft matter.
   * Modified Bleeding Index (mBI) (29)will be recorded at four aspects (mesial, distal, buccal, and lingual) around each implant at T3 and T4:

     * Score 0: No bleeding when a periodontal probe is passed along the mucosal margin adjacent to the implant.
     * Score 1: Isolated bleeding sport visible.
     * Score 2: Blood forms a confluent red line on mucosal margin.
     * Score 3: Heavy or profuse bleeding.
   * Width of keratinized tissue (KT) measured mid-facially from the gingival margin to the mucogingival junction of the intended extracted tooth (T0) or the implant-supported restoration (T3 and T4); or, from the top of edentulous crest to the mucogingival junction of the edentulous area (T1 and T2).
   * Facial soft tissue levels (STL) will be evaluated (at baseline (T0), and at T1, T2, T3, and T4) measuring the distance between level of soft tissues at mid-

   facial gingival level and a reference line, which connected the facial soft tissue level of the adjacent teeth.

   - Pink esthetic score (PES) will be evaluated at the end of the evaluation period. The PES is based in 7 variables: mesial papilla, distal papilla, soft tissue level, soft tissue contour, alveolar process deficiency, soft tissue color and soft tissue texture. Each variable will be assessed with a 2-1-0 score with 2 being the best and 0 being the worst score. The highest possible score reflecting a perfect match of the peri-implant soft tissue with that of the reference tooth is 14 and the lowest score reflecting a bad match of the peri-implant soft tissue is 0 (26).

   5.5.3 Intra-surgical parameters

   After tooth extraction, a periodontal probe PCP-UNC 15 (HuFriedy, Rockwell St, Chicago, IL) will be used to measure the vertical distance (VD) between the buccal gingival margin and the bone wall.

   5.5.4 Radiographic parameters

   A calibrated examiner (P.D.) will evaluate the following radiographic parameters:

   Horizontal measurements

   CBCT scans will be obtained at the time of tooth extraction (T0) and after 3 months (T1) (approximately 2 weeks before implant installation for treatment planning) and 12 months (T4). Width measurements will be performed to compare differences between groups after a healing period of 3 and 12 months. For each socket, a longitudinal (parallel to the root cross section) view will be obtained.

   According to Sisti et al. (22), the total width (TW) of the buccolingual bone will be measured at three horizontal lines perpendicular to the long axis of the post-extraction socket: 1 mm (total coronal width, TW1), 4 mm (total median width, TW4), and 7 mm apical to the palatal bone crest (total apical width, TW7). On the same lines, palatal bone wall (PW) will be also measured: coronal palatal width (PW1), median palatal width (PW4), and apical palatal width (PW7).

   Vertical measurements

   According to Araújo et al. (2), the VD between the palatal and buccal wall peaks will be measured in CBCT scans.

   Intra-oral periapical radiographs with a bite block will be taken with the long cone paralleling technique (7mA-60kV/20ms) at T1, T2, T3, and T4 (6 months after implant placement). A paralleling device and individualized bite blocks (Optosil) will be used for the standardisation of the X-ray geometry. The marginal bone height (MBL) will be set as the distance between the reference point and the most apical point of the marginal bone level. The reference point will be the fixture- abutment interface. Calibration will be performed using the known thread-pitch distance of the implants. Previously known values, such as mixture diameter and length, will be used for calibration when the threads will not be clearly visible on the radiographs. The digitally obtained X-rays will be transferred into a software program (Image J; NIH, Bethesda, MD, USA).

   CBCT analysis Along the 1 year protocol duration of the present investigation, three CBCT scan will be needed; At baseline, the first CBCT will be taken immediately following extraction in order to get accurate images of the ridge status. At 3 months, and before implant placement, a second CBCT scan will be taken, included in the implant study and it will be useful to compare with the initial CBCT analysis in both groups. Last of all, at 1 year follow-up a third CBCT scan will be taken in both groups; In the control group, it will be useful to make comparisons before and after bone graft over the implant, and in the test group it will allow to make comparisons with the control group about the buccal plate status.

   5.5.5 Volumetric analysis

   Alginate impressions will be taken at the baseline examination (T0), and at T1, T2, T3, and T4. Dental stone casts will be fabricated immediately after the impressions will be obtained. Models will be evaluated for the presence of irregularities such as porous areas, undefined gingival margins, broken cusps, or undefined vestibulum.

   The cast models will be optically scanned with a desktop 3D scanner. Baseline and follow-up STL files of the models will be uploaded to an image analysis software (Swissmeda Software; Swissmeda AG, Zurich, Switzerland). To match the STL files, three clear and visible common reference points will be selected. After the selection of these references, the software automatically superimposed the models using a series of mathematical algorithms. Linear and volumetric measurements will be performed by a calibrated evaluator.

   Stages of the volumetric analysis
   * Test group

     * Volume preservation: from T0 to T1
     * Volume stability: from T1 to T2
     * Volume gain (after SCTG): from T2 to T3
     * Volume stability: from T3 to T4
   * Control group:

     * Volume loss: from T0 to T1
     * Volume gain (after regenerative procedure): from T1 to T2
     * Volume gain (after SCTG): from T2 to T3
     * Volume stability: from T3 to T4

   5.5.6 Intra-examiner reproducibility

   The intra-examiner reliability will be estimated. The degree of intraobserver agreement of total width (TW) of the buccolingual bone (mm), measured in CBCT scans, will be determined with the Interclass Correlation Coefficient (ICC). All measurements will be taken by one examiner (P.D.).

   The examiner will be calibrated as follows, five patients not involved in the study with a CBCT scan will be recruited and used for calibration. The examiner will record the total width (TW) of the buccolingual bone (measured at three horizontal lines perpendicular to the long axis of the ridge: 1 mm, 4 mm, and 7 mm apical to the palatal

   bone crest) on two separate occasions 48 hours apart. Cali¬bration will be accepted if 90% of the recordings could be reproduced within a difference ≤ 0.1 mm.

   5.6 Outcomes
   * Primary outcome: Total width (TW) of the buccolingual bone measured in CBCT scans.
   * Secondary outcomes: KT, STL, PES, volumetric soft tissue changes, and radiographic bone loss.

   5.7 Withdrawal of consent

   The Patient Information Sheet will clearly state that the patient can withdraw from the study at any time without prejudice or explanation. Such withdrawal will be documented in the medical record file. Losses to follow-up are taken into account in the sample size calculations (12%).

   5.8 Sample size calculation

   Using the total width (W) of the buccolingual bone as the primary outcome variable, the sample size was calculated. Power calculation based on the detection of a clinically significant difference ≥ 3 mm in mean crest-dimension difference between treatment groups, assuming a standard deviation of 2.5 mm (Schropp et al. 2003), with an alpha error defined to 0.05 and beta error to 0.20 (power 80%), revealed that 12 subjects in each treatment group were required. In addition, an estimation that 20% of subjects will be lost to follow-up has been taken into account.
6. Result analysis:

6.9 Statistical analysis

The study variables will be recorded in a case report form (CRF) specially designed for the study. Each study patient will be assigned a numerical code comprising a 3-digit patient code (assigned correlatively as they are included in the study). Only the study investigator will be able to identify the patient by their code.

At the end of the fieldwork, the data contained in the CRFs will be entered into a database for data analysis and preparation of the final report.

The socio-demographic and clinical characteristics and other variables of interest of the patients included in the study will be described. Data will be presented as mean ± SD; categorical data will be shown as percentage of positive patients.

An analysis will be carried out to determine differences in study outcomes between groups. Analysis will be based on the ITT (intention to treat) population using the last observation carried forward (LOCF) approach. The relationship between two qualitative variables will be calculated using the chi-squared test or Fisher's exact test (if in a given case the frequency observed is < 5). For ordinal variables, linear regression will be calculated using Kendall's tau coefficient.

Quantitative variables will be compared using the Student's t-test (< 2 categories), analysis of variance [ANOVA] (for variables > 2 categories), linear regression test and Scheffé's multiple comparisons test or U Mann Whitney non-parametric test. The linear relationship between the quantitative variables will be calculated using Pearson's correlation coefficient or Spearman's rank correlation test (if the variable is not normally distributed). Changes vs. baseline will be analyzed using the Wilcoxon non-parametric test or Mc Nemar test.

Level of significance will be set at 0.05. The SPSS version 19.00 software (SPSS Inc., Chicago, IL, USA) will be used for all analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women over 18 years old.
2. Patients requiring single tooth extraction with partial or total absence of the buccal bone wall that will be defined as loss of more than 5 mm with respect to the supposed location of the bone crest (23).
3. Presence of adjacent teeth.
4. Anterior teeth (from second premolar to second premolar) of the maxilla.
5. Patients who had requested an implant restoration between adjacent teeth
6. Absence of active periodontal disease.
7. Good level of oral hygiene (Plaque Index < 25%; (27).
8. Absence of systemic diseases that could influence the outcome of the therapy (i.e. uncontrolled diabetes mellitus, osteoporosis, biphosphonate medication).
9. Non-smokers or light smokers (< 10 cigarettes per day).
10. Written informed consent signed.

Exclusion Criteria:

1. Buccal soft tissue recession.
2. Acute infection at the extraction site.
3. Presence of adjacent implants.
4. Absence of any adjacent tooth
5. Long-term non-steroidal anti-inflammatory drug therapy (3 months).
6. Lactating females or currently pregnancy.
7. Severe cognitive or psychiatric disorders.
8. Unwillingness to return for follow-up examination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-02 (Actual); Primary Completion 2018-11 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
total width of the buccolingual bone | Baseline, 3 months, 1 year
  to evaluate the bone changes in cone beam computed tomography

SECONDARY OUTCOMES:
keratinized tissue | Baseline, 3 months and at 1 year
  to evaluate the height of keratinized tissue in millimeters
soft tissue level | Baseline, 3 months and at 1 year
  to evaluate the recession of the gingiva in millimeters
pink esthetic score | Baseline, 3 months and at 1 year
  evaluate the final delivery prosthesis over implant
volumetric soft tissue changes (linear measurement) | At 3 months and at 1 year
  To compare soft tissue changes between baseline and follow ups measured in millimeters
radiographic bone loss (in millimeters) | At 3 months, and at 1 year
  changes in periapical radiographs measured in millimeters from the implant neck to the first bone to implant contact

CONTACTS AND LOCATIONS:
Overall Officials: PEDRO DIZ, Principal Investigator — Universitat Internacional de Catalunya
Locations (1):
- Universitat Internacional de Catalunya, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: Undecided